CLINICAL TRIAL: NCT02608242
Title: A Randomized, Open-label, Single Dose, Crossover Clinical Trial to Compare the Safety and Pharmacokinetics of YH22189 in Comparison to Telmisartan/Amlodipine and Rosuvastatin in Healthy Volunteers
Brief Title: PK Study of YH22189 FDC Compared to Combination of Telmisartan/Amlodipine and Rosuvastatin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH22189-102
Record Dates: First submitted 2015-11-11; First posted 2015-11-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — telmisartan amlodipine combination; Telmisartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- YH22189 (Experimental): YH22189 FDC tablet of Yuhan Corporation
  Interventions: Drug: YH22189
- Twynsta 80/10mg (Active Comparator): Telmisartan/Amlodipine 80/10mg (FDC)
  Interventions: Drug: Twynsta 80/10mg
- Crestor 20mg (Active Comparator): Rosuvastatin 20mg
  Interventions: Drug: Crestor 20mg

INTERVENTIONS:
Drug: YH22189
  Arms: YH22189
Drug: Twynsta 80/10mg
  Other Names: Telmisartan/Amlodipine 80/10mg(FDC)
  Arms: Twynsta 80/10mg
Drug: Crestor 20mg
  Other Names: Rosuvastatin 20mg
  Arms: Crestor 20mg

SUMMARY:
This is a Randomized, open-label, single-dose, 3-treatment, 3-period, 3-sequence crossover design.

DETAILED DESCRIPTION:
This is a 6 by 3 cross-over study to evaluate pharmacokinetics of YH22189 FDC compared to reference telmisartan/amlodipine and rosuvastatin co-administered in three groups enrolling healthy adult male subjects under fasting conditions.

Subjects will be admitted to the clinic in the evening before Day 1. All subjects will receive a single oral dose of YH22189 FDC or telmisartan/amlodipine or rosuvastatin administered in the morning on Day 1. All the subjects will remain in the clinical unit until completion of all assessments on Day 2 including collection post-dose PK sample. Subjects will return to the clinic for pharmacokinetic samples at scheduled time. The three treatment periods will be separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female with a body mass index(BMI) between 18.5 and 25 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
* Administration of other investigational products within 3 months prior to the first dosing
* Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs
* Sitting blood pressure meeting the following criteria at screening: 150 ≥ systolic blood pressure ≤100 (mmHg) and 100 ≥ diastolic blood pressure ≤ 60 (mmHg)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Telmisartan Cmax | 0 - 72 hrs
Telmisartan AUClast | 0 - 72 hrs
Amlodipine Cmax | 0 - 168 hrs
Amlodipine AUClast | 0 - 168 hrs
Rosuvastatin Cmax | 0 - 48 hrs
Rosuvastatin AUClast | 0 - 48 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No